CLINICAL TRIAL: NCT07399262
Title: Music-Augmented Versus Non-Music Technology-Based Rhythmic Gait Training in Multiple Sclerosis: A Randomized Controlled Trial of Gait Performance and Clinical Outcomes
Brief Title: Music-Augmented Rhythmic Gait Training in Multiple Sclerosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Guzin Kaya Aytutuldu, Assistant Professor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Biruni.U
Record Dates: First submitted 2026-01-29; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Multiple Sclerosis; Rehabilitation
Keywords: Multiple Sclerosis; Rhythmic Gait Training; Music-Based Exercise; Telerehabilitation; Gait Performance
MeSH Terms: conditions — Multiple Sclerosis | interventions — Respiration

STUDY DESIGN:
Intervention Model Description: This study is a two-arm, parallel-group, randomized controlled trial comparing music-assisted rhythmic gait training with non-music rhythmic gait training, conducted without masking due to the nature of the interventions.
Masking Description: This study is a two-arm, parallel-group, randomized controlled trial comparing music-assisted rhythmic gait training with non-music rhythmic gait training, conducted without masking due to the nature of the interventions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rhythmic GaitTraining Group with Music (Experimental): Participants in this group will perform technology-based rhythmic gait exercises accompanied by music. The intervention will be delivered via telerehabilitation under the supervision of a physiotherapist, four days per week for four weeks.
  Interventions: Other: Breathing and General Mobility Exercises; Other: Music-Assisted Rhythmic Gait Training
- Rhythmic Gait Training Without Music (Active Comparator): Participants in this group will perform the same technology-based rhythmic gait exercises without music. The intervention will be delivered via telerehabilitation under the supervision of a physiotherapist, four days per week for four weeks.
  Interventions: Other: Breathing and General Mobility Exercises; Other: Rhythmic Gait Training Without Music

INTERVENTIONS:
Other: Breathing and General Mobility Exercises — rticipants will perform standardized breathing exercises and general mobility exercises. These exercises will be delivered in the same telerehabilitation format and supervised by a physiotherapist.
Other: Music-Assisted Rhythmic Gait Training — Participants will perform rhythmic gait training accompanied by music. The training will be delivered via telerehabilitation with real-time supervision through videoconferencing. Sessions will be conducted four days per week for four weeks. Gait training will be guided using instructional videos presented with music accompaniment.
  Arms: Rhythmic GaitTraining Group with Music
Other: Rhythmic Gait Training Without Music — Participants will perform the same rhythmic gait training program without music. The training will be delivered via telerehabilitation with real-time supervision through videoconferencing. Sessions will be conducted four days per week for four weeks. Gait training will be guided using instructional videos presented without music (silent).
  Arms: Rhythmic Gait Training Without Music

SUMMARY:
This randomized controlled trial aims to compare the effects of technology-based rhythmic gait training performed with and without music on walking performance and clinical outcomes in individuals with multiple sclerosis (MS). Thirty-two participants with mild to moderate disability will be randomly assigned to either a music-assisted rhythmic gait training group or a non-music control group, with both interventions delivered via telerehabilitation. Outcomes related to gait performance, balance, fatigue, and cognitive function will be assessed before and after a four-week intervention period.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic, inflammatory, and demyelinating disease of the central nervous system that leads to impairments in motor and cognitive functions, with gait disturbances being among the most common and disabling symptoms. Walking impairments in individuals with MS substantially reduce quality of life and are frequently accompanied by balance deficits, fatigue, and decreased functional capacity, ultimately limiting independence in daily activities.

Recent evidence suggests that rhythmic auditory stimulation and music-based gait training can enhance motor control and walking performance by providing external temporal cues that facilitate movement coordination. In parallel, telerehabilitation has emerged as an effective and accessible rehabilitation approach, enabling supervised exercise delivery while reducing barriers related to transportation, cost, and long-term adherence.

In this randomized controlled trial, a total of 32 individuals with MS who have an Expanded Disability Status Scale (EDSS) score between 0 and 4 and a definite diagnosis according to the McDonald criteria will be recruited. Participants will be randomly allocated into two groups using computer-generated randomization. The intervention group (Group A) will perform rhythmic gait exercises accompanied by music, whereas the control group (Group B) will perform the same exercises without music. Both interventions will be delivered in a telerehabilitation format under the supervision of a physiotherapist.

The intervention program will last four weeks, with training sessions conducted four days per week. Primary and secondary outcome measures assessing walking performance, balance, fatigue, and cognitive function will be administered before and after the intervention period.

The primary objective of this study is to comparatively evaluate the effects of technology-based, music-assisted rhythmic gait training on motor outcomes in individuals with MS and to contribute high-quality scientific evidence to an area that remains underrepresented in the current rehabilitation literature.

ELIGIBILITY:
Inclusion Criteria:

* Expanded Disability Status Scale (EDSS) score between 0 and 4.0

Access to the internet via a high-speed smartphone or computer

A score of at least 21 on the Montreal Cognitive Assessment (MoCA)

Functional Ambulation Scale score of Stage 3 or higher

Exclusion Criteria:

* Presence of hearing or visual impairments

Current participation in any structured exercise program

Presence of other neurological, cardiovascular, or orthopedic disorders

History of MS relapse or change in disease-modifying treatment within the last 6 months

Physical conditions preventing safe participation in the exercise program

Comorbid conditions that adversely affect oxygen transport (e.g., severe anemia, peripheral arterial disease)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Gait Speed | Baseline and immediately after intervention
  Walking speed is the primary outcome measure of the study and will be assessed using the Timed 25-Foot Walk Test (T25FW). In this test, participants are instructed to walk a distance of 7.62 m (25 feet) as quickly and safely as possible, without running. The completion time is recorded in seconds. Two trials are performed, and the average of the two trials is recorded as the T25FW score. The T25FW is one of the most well-established and widely used measures for assessing gait impairment and walking speed in individuals with multiple sclerosis

SECONDARY OUTCOMES:
Two Minute Walk Test | Baseline and immediately after intervention
  The Two-Minute Walk Test (2MWT) will be used to assess functional walking capacity and treatment response. The total distance walked within two minutes is recorded in meters. Vital signs are measured before and after the test. In this study, the 2MWT is preferred over the 6-Minute Walk Test due to its practicality, feasibility, and validated use in individuals with MS without inducing excessive fatigue
Timed Up and Go Test | Baseline and immediately after intervention
  In the Timed Up and Go Test, participants are instructed to stand up from a seated position, walk a distance of 3 meters, turn around a reference object, return to the chair, and sit down. The time required to complete the task is recorded in seconds. The test is performed three times, and the average time is used for analysis
Step Length | Baseline and immediately after intervention
  Kinovea® software (version 0.8.15) is used to perform objective and quantitative kinematic and spatiotemporal gait analysis from video recordings. The software enables the analysis of parameters such as step length, stride length, base of support, step width, cadence, walking speed, and step time (37).
  In this study, gait will be recorded using a camera positioned in the sagittal plane while participants walk a distance of 3 meters. Colored markers will be placed on the right and left heels to facilitate identification in the video recordings. Several gait cycles will be captured and analyzed independently using Kinovea software to determine step length (distance between consecutive heel strikes of opposite limbs), stride length (distance between consecutive heel strikes of the same limb), cadence (steps per minute), and bilateral step lengths (38-40). Walking speed (V) will be calculated using the formula:
Stride Length | Baseline and immediately after intervention
  Kinovea® software (version 0.8.15) is used to perform objective and quantitative kinematic and spatiotemporal gait analysis from video recordings. The software enables the analysis of parameters such as step length, stride length, base of support, step width, cadence, walking speed, and step time (37).
  In this study, gait will be recorded using a camera positioned in the sagittal plane while participants walk a distance of 3 meters. Colored markers will be placed on the right and left heels to facilitate identification in the video recordings. Several gait cycles will be captured and analyzed independently using Kinovea software to determine step length (distance between consecutive heel strikes of opposite limbs), stride length (distance between consecutive heel strikes of the same limb), cadence (steps per minute), and bilateral step lengths (38-40). Walking speed (V) will be calculated using the formula:
Walking Speed | Baseline and immediately after intervention
  Kinovea® software (version 0.8.15) is used to perform objective and quantitative kinematic and spatiotemporal gait analysis from video recordings. The software enables the analysis of parameters such as step length, stride length, base of support, step width, cadence, walking speed, and step time (37).
  In this study, gait will be recorded using a camera positioned in the sagittal plane while participants walk a distance of 3 meters. Colored markers will be placed on the right and left heels to facilitate identification in the video recordings. Several gait cycles will be captured and analyzed independently using Kinovea software to determine step length (distance between consecutive heel strikes of opposite limbs), stride length (distance between consecutive heel strikes of the same limb), cadence (steps per minute), and bilateral step lengths (38-40). Walking speed (V) will be calculated using the formula:
Modified Fatigue Impact Scale | Baseline and immediately after intervention
  The Modified Fatigue Impact Scale (MFIS) is a 21-item questionnaire designed to assess the impact of fatigue on physical, cognitive, and psychosocial functioning (41). Each item is scored on a 5-point Likert scale ranging from 0 (no problem) to 4 (severe problem). The total score ranges from 0 to 84, with higher scores indicating greater fatigue severity. Subscale scores for physical, cognitive, and psychosocial domains are calculated and summed to obtain the total score.
The Four Square Step Test | Baseline and immediately after intervention
  The Four Square Step Test evaluates the ability to change direction while stepping. Participants begin in Square 1 (upper left) and follow a predefined stepping sequence clockwise (Squares 1-2-4-3) and then counterclockwise (Squares 3-4-2-1). The physiotherapist demonstrates the test and allows practice trials if needed. If the participant loses balance, touches the assistive device, or fails to complete the sequence, the test is repeated. Two trials are recorded, and the best performance time is used for analysis. Timing begins when the first foot contacts Square 2 and ends when both feet return to Square 1
BICAMS Battery | Baseline and immediately after intervention
  The BICAMS battery includes the Symbol Digit Modalities Test (SDMT), California Verbal Learning Test-Second Edition (CVLT-II), and Brief Visuospatial Memory Test-Revised (BVMT-R). The battery was recommended in 2012 for monitoring cognitive function in individuals with MS, and its Turkish validity and reliability were established in 2017

CONTACTS AND LOCATIONS:
Overall Officials: Guzin Kaya Aytutuldu, Principal Investigator — Biruni University
Locations (1):
- Biruni University, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benedetti MG, Piperno R, Simoncini L, Bonato P, Tonini A, Giannini S. Gait abnormalities in minimally impaired multiple sclerosis patients. Mult Scler. 1999 Oct;5(5):363-8. doi: 10.1177/135245859900500510. PMID 10516781
- [Background] Ehde DM, Elzea JL, Verrall AM, Gibbons LE, Smith AE, Amtmann D. Efficacy of a Telephone-Delivered Self-Management Intervention for Persons With Multiple Sclerosis: A Randomized Controlled Trial With a One-Year Follow-Up. Arch Phys Med Rehabil. 2015 Nov;96(11):1945-58.e2. doi: 10.1016/j.apmr.2015.07.015. Epub 2015 Aug 6. PMID 26254948
- [Background] Conklyn D, Stough D, Novak E, Paczak S, Chemali K, Bethoux F. A home-based walking program using rhythmic auditory stimulation improves gait performance in patients with multiple sclerosis: a pilot study. Neurorehabil Neural Repair. 2010 Nov-Dec;24(9):835-42. doi: 10.1177/1545968310372139. Epub 2010 Jul 19. PMID 20643882